CLINICAL TRIAL: NCT03389035
Title: Phase 1-2a Trial to Determine the Feasibility and Safety of a Single Dose of Transposon-manipulated Allogeneic CARCIK-CD19 Cells in Adult and Pediatric Patients With Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia, After Hematopoietic Stem Cell Transplantation
Brief Title: Transposon-manipulated Allogeneic CARCIK-CD19 Cells in Pediatric and Adult Patients With r/r ALL Post HSCT
Acronym: CARCIK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Matilde Tettamanti Menotti De Marchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT01CARCIK
Record Dates: First submitted 2017-12-24; First posted 2018-01-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse
Keywords: Acute Lymphoblastic Leukemia; CAR-T; CARCIK; Transposon
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARCIK-CD19 (Experimental)
  Interventions: Biological: CARCIK-CD19

INTERVENTIONS:
Biological: CARCIK-CD19 — Allogeneic (donor-derived) Cytokine Induced Killer (CIK) cells transduced with a transposon CD19 Chimeric Antigen Receptor (CAR) gene

SUMMARY:
This is a single arm, open-label, multi-center, phase 1-2a study to determine the Maximum Tolerated Dose and/or the Recommended Phase 2 Dose and the safety of CARCIK-CD19 in adult and pediatric patients with relapsed or refractory B-cell precursor acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Children (1-17) and adults (18-75 years old);
* Relapsed or refractory adult and pediatric B-cell precursor ALL after HSCT;
* Evidence of CD19 tumor expression in bone marrow and/or peripheral blood by flow cytometry;
* Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening;
* No evidence of overall aGVHD > Grade I or chronic GVHD (cGVHD) greater than mild at time of enrollment and in the previous 30 days;
* No longer taking immunosuppressive agents for at least 30 days prior to enrollment;

Exclusion Criteria:

* Patients with GVHD Grades II-IV;
* Any cell therapy in the last 30 days;

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT): | 1 month
  rate and severity of the cytokine release syndrome (CRS)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale PG23, Bergamo, BG
  - Fondazione MBBM, Monza, MB

REFERENCES:
- [Derived] Magnani CF, Gaipa G, Lussana F, Belotti D, Gritti G, Napolitano S, Matera G, Cabiati B, Buracchi C, Borleri G, Fazio G, Zaninelli S, Tettamanti S, Cesana S, Colombo V, Quaroni M, Cazzaniga G, Rovelli A, Biagi E, Galimberti S, Calabria A, Benedicenti F, Montini E, Ferrari S, Introna M, Balduzzi A, Valsecchi MG, Dastoli G, Rambaldi A, Biondi A. Sleeping Beauty-engineered CAR T cells achieve antileukemic activity without severe toxicities. J Clin Invest. 2020 Nov 2;130(11):6021-6033. doi: 10.1172/JCI138473. PMID 32780725